CLINICAL TRIAL: NCT04287088
Title: Prebiopsy Magnetic Resonance Imaging in Men With Suspicion of Prostate Cancer - A Multi-centre Trial on Clinical Utility of IMPROD bpMRI in a Shared Decision Making Setting
Brief Title: bpMRI and Risk Based Shared Clinical Decision Making in Prostate Cancer Diagnosis
Acronym: multiIMPROD2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Tampere University Hospital (Other); Satakunta Central Hospital (Other); Central Finland Hospital District (Other); Memorial Sloan Kettering Cancer Center (Other); Mount Sinai Hospital, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: T326/2019
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Prostate Cancer
Keywords: bpMRI; shared decision making; IMPROD; risk calculation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): After IMPROD bpMRI all men undergo prostate biopsies. In men with Likert scores of 1-2, TRUS guided systematic biopsies are performed. In men with Likert 3-5 score, in addition to systematic biopsies, two targeted biopsies are taken from each lesion (up to two lesions).
- Intervention (Experimental): After IMPROD bpMRI prostate biopsies are performed according to shared decision-making by the treating urologist and the patient. If biopsies are to be performed, in men with IMPROD bpMRI likert scores of 1-2, 12-core systematic TRUS guided biopsies are performed and in men with Likert 3-5 score lesions systematic biopsies are performed and two targeted biopsies are taken from each lesion (up to two lesions). If biopsies are not performed, men are referred for a PSA follow-up.
  Interventions: Diagnostic Test: A shared decision making

INTERVENTIONS:
Diagnostic Test: A shared decision making — Based on prostate cancer risk calculation (age, usage of 5-ARI medication, baseline PSA, IMPROD bpMRI Likert, prostate volume) a shared decision making whether to perform prostate biopsies or not
  Arms: Intervention

SUMMARY:
The shortcoming of the pre-biopsy prostate MRI approach is the recommendation to biopsy all men post-MRI even if there is no lesion seen in MRI, ie. risk of PCa is very low. Therefore, the primary objective of this trial is to compare if there is a difference between significant cancer detection rate in men undergoing prostate biopsies after MRI scan compared to men undergoing post-MRI prostate biopsies only after a shared decision-making based on prostate cancer risk estimation.

The trial will enrol 600 patients. The primary outcome measure is the the proportion of men with CSPCa (Gleason 4+3 prostate cancer or higher) between the control and intervention arms at baseline. Eligible men are randomised 1:1 in two groups. In control arm in all men prostate biopsies are performed after MRI whereas in intervention arm prostate biopsies are performed only after a shared decision-making between urologist and the patient and the discussion is based on risk estimation.

DETAILED DESCRIPTION:
Although most of the prostate cancers (PCas) are currently being diagnosed at early stage, at present, 30% of men are diagnosed with primarily metastatic disease. The need for better diagnostic methods is, therefore, warranted. Recent studies have shown that an alternative pathway using multiparametric (mpMRI) or biparametric (bpMRI) magnetic resonance imaging as a triage test reduces unnecessary biopsies, decreases the detection of clinically non-significant PCa (non-SPCa), and improves the detection of clinically significant PCa (CSPCa). In addition, based on these trials, also EAU guideline was updated to recommend that all men should undergo pre-biopsy mpMRI. However, shortcoming of the approach is the recommendation to biopsy all men post-MRI even if there is no lesion seen in MRI, ie. risk of PCa is very low. Therefore, the primary objective of this randomised controlled trial is to compare if there is a difference between significant cancer detection rate in men undergoing prostate biopsies after MRI scan compared to men undergoing post-MRI prostate biopsies only after a shared decision-making based on prostate cancer risk estimation.

The trial will enrol 600 patients from four hospital districts: Varsinais-Suomi, Satakunta, Pirkanmaa and Keski-Suomi. Key inclusion criteria are suspicion of prostate cancer based on elevated PSA and/or abnormal digital rectal examination. Men with previous PCa diagnosis and contraindications for MRI are excluded. The primary outcome measure is the comparison of the proportion of men with CSPCa (Gleason 4+3 prostate cancer or higher) between the control and intervention arms at baseline.

Using PSA as strata, eligible men are randomised 1:1 in two groups. After randomisation MRI examination is performed and interpreted by one experienced uro-radiologist using Likert and PI-RADS2.1 classifications. In control arm in all men prostate biopsies are performed after MRI whereas in intervention arm prostate biopsies are performed only after a shared decision-making between urologist and the patient and the discussion is based on risk estimation. Men with negative biopsies or with no biopsies performed are all assigned for five-year follow-up with semi-annual PSA. Long-term follow-up based on health records and national registries is performed for additional 15 years for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Language spoken: Finnish
* Clinical suspicion of prostate cancer, based on: serum level of PSA from 2,5 ng/ml to 20 ng/ml and/or abnormal digital rectal examination according to the referral physician
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* previous diagnosis of prostate cancer
* any contraindications for MRI
* any other conditions that might compromise patient's safety, based on the clinical judgment of the responsible urologist
* bilateral hip prosthesis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Gleason 4+3=7 prostate cancer, baseline | baseline
  The proportion of men with clinically significant prostate cancer (Gleason 4+3 [ISUP grade group, the GGG, 3]) prostate cancer or higher) in the control and intervention arms after primary diagnostic pathway

SECONDARY OUTCOMES:
Gleason 3+4=7 or lower prostate cancer, baseline | baseline
  The proportion of men with clinically non-significant prostate cancer and intermediate risk prostate cancer (Gleason 3+3 [GGG 1], and Gleason 3+4 [GGG 2]) and benign biopsies in the control and intervention arms after primary diagnostic pathway
Men undergoing biopsies | baseline
  The proportion of men undergoing biopsies in the control and intervention arms
Biopsy related complications | baseline
  The proportion of men having biopsy-related complications in the control and intervention arms
Gleason 4+3=7 prostate cancer, follow-up | during the five years of follow-up
  The proportion of men with clinically significant prostate cancer (Gleason 4+3 [GGG 3], prostate cancer or higher) in the control and intervention arms during the five years of follow-up
the Memorial Anxiety Scale for Prostate Cancer -questionnaire (MAX-PC) | baseline, 6months, 12months
  Total score in MAX-PC in the control and intervention arms. Score range: 0-54. Higher scores in MAX-PC denote higher anxiety.
Biopsy probability | baseline
  The probability of performing biopsy in experimental arm

OTHER OUTCOMES:
Biopsy criteria outcome | baseline
  The number of biopsies and the number of clinically significant prostate cancer detected for each biopsy criteria
Calibration of the model | Baseline
  Calibration of the model using both Likert and PI-RADS2.1 criteria
Calibration of the model using biomarkers | Baseline
  Calibration of the model using biomarkers such as the four kallikrein panel

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Central Finland Central Hospital, Jyväskylä
  - Satakunta Central Hospital, Pori
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be published in peer-reviewed journal. Also, all MRI scans (pseudoanonymised), MRI reports, calculator risk scores and relevant clinical data will be provided online and publicly available similarly to previous IMPROD studies, see Links below. Informed consent form and analytic code are shared upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and SAP will be published during spring 2020. MRI scans, MRI reports, calculator risk scores and clinical data will be published at the time of the actual publication.
Access Criteria: Publicly available. Free access.

REFERENCES:
- [Derived] Ettala O, Jambor I, Montoya Perez I, Seppanen M, Kaipia A, Seikkula H, Syvanen KT, Taimen P, Verho J, Steiner A, Saunavaara J, Saukko E, Loyttyniemi E, Sjoberg DD, Vickers A, Aronen H, Bostrom P. Individualised non-contrast MRI-based risk estimation and shared decision-making in men with a suspicion of prostate cancer: protocol for multicentre randomised controlled trial (multi-IMPROD V.2.0). BMJ Open. 2022 Apr 15;12(4):e053118. doi: 10.1136/bmjopen-2021-053118. PMID 35428621
- See also: multi-IMPROD trial — http://petiv.utu.fi/multiimprod
- See also: IMPROD trial — http://petiv.utu.fi/improd/